CLINICAL TRIAL: NCT06711549
Title: "Serratus Anterior Plane Block" Versus "Serratus Posterior Superior Plane Intercostal Plane Block" for Patients Undergoing Breast Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale di Camposampiero (Other)
Collaborators: Azienda Ulss 6 Euganea (Other)
Responsible Party: Principal Investigator, Valentina Scaduto, Medical Doctor, Ospedale di Camposampiero
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/Sapvsspis
Record Dates: First submitted 2024-10-20; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Pain, Postoperative; Breast Cancer; Anesthesia; Mastectomy
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients receiving Serratus Posterior Superior Plane Intercostal Plane block (Experimental): The patients will undergosurgery after receiving an ultrasound guided serratus posterior superior intercostal plane block
  Interventions: Procedure: Serratus Posterior Superior Plane Intercostal Plane block
- Serratus Anterior Plane Block (Active Comparator): The patients will undergosurgery after receiving an ultrasound guided serratus anterior plane block
  Interventions: Procedure: Serratus Anterior Plane block

INTERVENTIONS:
Procedure: Serratus Posterior Superior Plane Intercostal Plane block — Under ultrasound guidance; local anesthetic will be injected in the plane between the posterior aspect of the serratus posterior superior plane and the ribs
  Arms: Patients receiving Serratus Posterior Superior Plane Intercostal Plane block
Procedure: Serratus Anterior Plane block — Under ultrasound guidance; local anesthetic will be injected in the plane between the posterior aspect of the serratus anterior and the external intercostal muscles and ribs
  Arms: Serratus Anterior Plane Block

SUMMARY:
The Serrato Posterosuperior Block (SPSIP) is a recently discovered technique that provides analgesia to the hemithorax, shoulders, neck and back. At an anatomical level, it has been seen that this technique allows the diffusion of local anesthetic starting from C7 proceeding dorsally up to T10 by sectioning the trapezius, latissimus dorsi, rhomboid and erector spinae muscles. The serratus anterior block (SAPB) is a technique that allows local anesthetic to be injected between the serratus anterior muscle and the intercostal muscles (deep plane) or between the latissimus dorsi muscle and the serratus anterior muscle (superficial plane), also providing analgesia at of the chest wall. This study aims to compare the analgesic efficacy of SPSIPB and SAPB in patients undergoing radical mastectomy for breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient ( > 18 years)
* Informed consent
* American Society of Anaesthesiologis Phisical Status I to III
* Patients undergoing for mastectomy with sentinel lynphnode byopsy/axillary clearence

Exclusion Criteria:

* Pregnant women
* Allergy to any drug present in the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain at 0 hours after surgery | 0 hours after surgery
  The primary objective of the study is to evaluate whether there is a difference between SAP block and SPSIP block at 0 hours after surgery at rest measure with visual analogic scale (0-10)

SECONDARY OUTCOMES:
Pain at 6 hours after surgery | 6 hours after surgery
  Evaluate whether there is a difference between SAP block and SPSIP block at 6 hours after surgery at rest measure with visual analogic scale (0-10)
Pain at 12 hours after surgery | 12 hours after surgery
  Evaluate whether there is a difference between SAP block and SPSIP block at 12 hours after surgery at rest measure with visual analogic scale (0-10)
Pain at 24hours after surgery | 24 hours after surgery
  Evaluate whether there is a difference between SAP block and SPSIP block at 24 hours after surgery at rest measure with visual analogic scale (0-10)
Intraoperative Opioid consumption | During the surgery(From patient intubation to patient extubation)
  Intraoperative opioids consumption (remifentanyl measured as mcg/kg)
Postoperative Opioid consumption | From extubation to 24 hours post-enrollment
  Postoperative use of rescue analgesics (measured as yes or no)
Postoperative Nausea and Vomiting | From extubation to 24 hours post-enrollment
  Postoperative Nausea and Vomiting defined as patient reporting nausea and vomiting or requiring drugs for nausea or vomiting

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rogobete AF, Sandesc D. General Anesthesia as a Multimodal Individualized Clinical Concept. Medicina (Kaunas). 2022 Jul 19;58(7):956. doi: 10.3390/medicina58070956. PMID 35888675
- [Result] Nelson G, Fotopoulou C, Taylor J, Glaser G, Bakkum-Gamez J, Meyer LA, Stone R, Mena G, Elias KM, Altman AD, Bisch SP, Ramirez PT, Dowdy SC. Enhanced recovery after surgery (ERAS(R)) society guidelines for gynecologic oncology: Addressing implementation challenges - 2023 update. Gynecol Oncol. 2023 Jun;173:58-67. doi: 10.1016/j.ygyno.2023.04.009. Epub 2023 Apr 21. PMID 37086524